CLINICAL TRIAL: NCT05655000
Title: A First-in-Humans Supermicrosurgical Technique for the Neonatal Thymus Transplantation
Brief Title: Neonatal Thymus Transplantation in Humans
Acronym: SUPERTHYM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FVL-1995
Record Dates: First submitted 2022-11-24; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Safety Issues
Keywords: Neonatal thymus transplant; First-in-humans; Clinical trial; Safety; Supermicrosurgery

STUDY DESIGN:
Intervention Model Description: Single-subject study of a supermicrosurgical technique for neonatal thymus transplantation in an adult with acute myeloid leukemia who is not candidate for bone marrow transplant, nor intensive chemotherapy. The participant will receive multidisciplinary supportive care before, during and after the procedure. The safety and adverse event profile will be assessed throughout the study. The graft will be explanted 14-21 days after the procedure. Thymopoiesis will be measured at baseline and at postoperatve day 14-21, before explantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonatal thymus transplantation (Experimental): Supermicrosurgical technique for neonatal thymus transplantation into the subject's radial forearm. The donor will be a neonate subject to corrective heart surgery via sternotomy requiring routinary partial thymectomy.
  Interventions: Procedure: Neonatal thymus transplantation

INTERVENTIONS:
Procedure: Neonatal thymus transplantation — The donor's neonatal thymus vessels will be dissected right after the routinary partial thymectomy. These vessels will be anastomosed into the recipient's penetrating vessels within the radial forearm by using a supermicrosurgical technique. The graft will be explanted at day 14-21 after the procedure.
  Other Names: Multidisciplinary supportive care before, during and after the procedure.

SUMMARY:
The goal of this clinical trial is to demonstrate the safety of the neonatal thymus transplant in an adult patient. The main questions it aims to answer are:

* Is the neonatal thymus transplant a safe procedure?
* What is the adverse event profile of the neonatal thymus transplant?

This is a single-subject study; thus, there will not be comparison groups. The participant will receive multidisciplinary supportive care before, during, and after the procedure.

DETAILED DESCRIPTION:
Inadequate thymopoiesis is probably related to autoimmunity, immunodeficiency, and immunosenescence. Enhancing thymopoiesis may be attractive for managing or studying such immunologic phenomena. Thymopoiesis is supported by the adult thymus transplant, as demonstrated in different animal models. Several approaches to enhance thymopoiesis in humans have been reported, which include in-vitro and in-vivo regeneration of the thymus and avascular grafting of allogeneic processed thymic tissue, among others.

Although a supermicrosurgical technique for neonatal thymus transplantation was recently described in rabbits, it has never been described in humans. This technique can be used to perform a neonatal thymus transplantation in humans. If this technique demonstrates to be safe, future studies will follow to investigate its effect on thymopoiesis and its efficacy on different health conditions.

This single-subject, first-in-humans clinical trial aims to demonstrate the safety and investigate the adverse effect profile of the neonatal thymus transplant in an adult with acute myeloid leukemia who is not candidate for bone marrow transplant, nor intensive chemotherapy. This human model not only allows to study the safety of the neonatal thymus transplant, it will also allow to investigate the effect of the procedure on thymopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute leukemia in palliative care, either myeloid (AML) or lymphocytic (ALL).
* Not candidate for bone marrow transplant.
* Not candidate for intensive chemotherapy.

Exclusion Criteria:

* Past medical history of bone marrow transplant.
* Past medical history of severe cognitive decline or dementia.
* Past medical history of severe liver failure.
* Past medical history of chronic kidney disease (CKD) stage 4-5.
* Past medical history of acute coronary syndrome within the past 90 days.
* Past medical history of acute ischemic stroke within the past 90 days.
* Past medical history of decompensated congestive heart failure (CHF) within the past 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 14-21 days
  Incidence of AEs and of clinically relevant changes in vital signs values, symptoms, physical examination findings, laboratory and imaging safety data.

SECONDARY OUTCOMES:
Thymic graft functioning | 14-21 days
  Change in percentage (%) of naïve (CD45+ CD3+ CDRA+) and memory (CD45+ CD3+ CDRA-) T lymphocytes over the total number of T lymphocytes by flow cytometry before engrafting (day -1), and before explant (day +14-21), as biomarkers of thymopoiesis.
Tissue viability | 14-21 days
  Presence and extent (if any) of the graft rejection by light microscopy with eosin-hematoxylin and immunochemistry staining in the explanted thymic tissue at post-operative day 14-21.
Donor-receptor compatibility | 14-21 days
  Human Leukocyte Antigens (HLA) typing.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Tintinago-Londoño, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle Del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bluestone JA, Anderson M. Tolerance in the Age of Immunotherapy. N Engl J Med. 2020 Sep 17;383(12):1156-1166. doi: 10.1056/NEJMra1911109. No abstract available. PMID 32937048
- [Background] Collins C, Sharpe E, Silber A, Kulke S, Hsieh EWY. Congenital Athymia: Genetic Etiologies, Clinical Manifestations, Diagnosis, and Treatment. J Clin Immunol. 2021 Jul;41(5):881-895. doi: 10.1007/s10875-021-01059-7. Epub 2021 May 13. PMID 33987750
- [Background] Mittelbrunn M, Kroemer G. Hallmarks of T cell aging. Nat Immunol. 2021 Jun;22(6):687-698. doi: 10.1038/s41590-021-00927-z. Epub 2021 May 13. PMID 33986548
- [Background] Bredenkamp N, Ulyanchenko S, O'Neill KE, Manley NR, Vaidya HJ, Blackburn CC. An organized and functional thymus generated from FOXN1-reprogrammed fibroblasts. Nat Cell Biol. 2014 Sep;16(9):902-8. doi: 10.1038/ncb3023. Epub 2014 Aug 24. PMID 25150981
- [Background] Velardi E, Tsai JJ, Holland AM, Wertheimer T, Yu VW, Zakrzewski JL, Tuckett AZ, Singer NV, West ML, Smith OM, Young LF, Kreines FM, Levy ER, Boyd RL, Scadden DT, Dudakov JA, van den Brink MR. Sex steroid blockade enhances thymopoiesis by modulating Notch signaling. J Exp Med. 2014 Nov 17;211(12):2341-9. doi: 10.1084/jem.20131289. Epub 2014 Oct 20. PMID 25332287
- [Background] O'Neill KE, Bredenkamp N, Tischner C, Vaidya HJ, Stenhouse FH, Peddie CD, Nowell CS, Gaskell T, Blackburn CC. Foxn1 Is Dynamically Regulated in Thymic Epithelial Cells during Embryogenesis and at the Onset of Thymic Involution. PLoS One. 2016 Mar 16;11(3):e0151666. doi: 10.1371/journal.pone.0151666. eCollection 2016. PMID 26983083
- [Background] Ulyanchenko S, O'Neill KE, Medley T, Farley AM, Vaidya HJ, Cook AM, Blair NF, Blackburn CC. Identification of a Bipotent Epithelial Progenitor Population in the Adult Thymus. Cell Rep. 2016 Mar 29;14(12):2819-32. doi: 10.1016/j.celrep.2016.02.080. Epub 2016 Mar 17. PMID 26997270
- [Background] Martin-Gayo E, Gonzalez-Garcia S, Garcia-Leon MJ, Murcia-Ceballos A, Alcain J, Garcia-Peydro M, Allende L, de Andres B, Gaspar ML, Toribio ML. Spatially restricted JAG1-Notch signaling in human thymus provides suitable DC developmental niches. J Exp Med. 2017 Nov 6;214(11):3361-3379. doi: 10.1084/jem.20161564. Epub 2017 Sep 25. PMID 28947612
- [Background] Shichkin VP, Gorbach OI, Zuieva OA, Grabchenko NI, Aksyonova IA, Todurov BM. Effect of cryopreservation on viability and growth efficiency of stromal-epithelial cells derived from neonatal human thymus. Cryobiology. 2017 Oct;78:70-79. doi: 10.1016/j.cryobiol.2017.06.010. Epub 2017 Jun 28. PMID 28668447
- [Background] Garcia-Leon MJ, Fuentes P, de la Pompa JL, Toribio ML. Dynamic regulation of NOTCH1 activation and Notch ligand expression in human thymus development. Development. 2018 Aug 13;145(16):dev165597. doi: 10.1242/dev.165597. PMID 30042180
- [Background] Campinoti S, Gjinovci A, Ragazzini R, Zanieri L, Ariza-McNaughton L, Catucci M, Boeing S, Park JE, Hutchinson JC, Munoz-Ruiz M, Manti PG, Vozza G, Villa CE, Phylactopoulos DE, Maurer C, Testa G, Stauss HJ, Teichmann SA, Sebire NJ, Hayday AC, Bonnet D, Bonfanti P. Reconstitution of a functional human thymus by postnatal stromal progenitor cells and natural whole-organ scaffolds. Nat Commun. 2020 Dec 11;11(1):6372. doi: 10.1038/s41467-020-20082-7. PMID 33311516
- [Background] Fahy GM. Apparent induction of partial thymic regeneration in a normal human subject: a case report. J Anti Aging Med. 2003;6(3):219-27. doi: 10.1089/109454503322733063. PMID 14987435
- [Background] Fahy GM, Brooke RT, Watson JP, Good Z, Vasanawala SS, Maecker H, Leipold MD, Lin DTS, Kobor MS, Horvath S. Reversal of epigenetic aging and immunosenescent trends in humans. Aging Cell. 2019 Dec;18(6):e13028. doi: 10.1111/acel.13028. Epub 2019 Sep 8. PMID 31496122
- [Background] Kirkpatrick JA Jr, DiGeorge AM. Congenital absence of the thymus. Am J Roentgenol Radium Ther Nucl Med. 1968 May;103(1):32-7. doi: 10.2214/ajr.103.1.32. No abstract available. PMID 5648947
- [Background] Conley ME, Beckwith JB, Mancer JF, Tenckhoff L. The spectrum of the DiGeorge syndrome. J Pediatr. 1979 Jun;94(6):883-90. doi: 10.1016/s0022-3476(79)80207-3. PMID 448529
- [Background] Thomas RA, Landing BH, Wells TR. Embryologic and other developmental considerations of thirty-eight possible variants of the DiGeorge anomaly. Am J Med Genet Suppl. 1987;3:43-66. doi: 10.1002/ajmg.1320280508. PMID 3130877
- [Background] Frank J, Pignata C, Panteleyev AA, Prowse DM, Baden H, Weiner L, Gaetaniello L, Ahmad W, Pozzi N, Cserhalmi-Friedman PB, Aita VM, Uyttendaele H, Gordon D, Ott J, Brissette JL, Christiano AM. Exposing the human nude phenotype. Nature. 1999 Apr 8;398(6727):473-4. doi: 10.1038/18997. No abstract available. PMID 10206641
- [Background] Pignata C, Fiore M, Guzzetta V, Castaldo A, Sebastio G, Porta F, Guarino A. Congenital Alopecia and nail dystrophy associated with severe functional T-cell immunodeficiency in two sibs. Am J Med Genet. 1996 Oct 16;65(2):167-70. doi: 10.1002/(SICI)1096-8628(19961016)65:23.0.CO;2-O. PMID 8911612
- [Background] Markert ML, Boeck A, Hale LP, Kloster AL, McLaughlin TM, Batchvarova MN, Douek DC, Koup RA, Kostyu DD, Ward FE, Rice HE, Mahaffey SM, Schiff SE, Buckley RH, Haynes BF. Transplantation of thymus tissue in complete DiGeorge syndrome. N Engl J Med. 1999 Oct 14;341(16):1180-9. doi: 10.1056/NEJM199910143411603. PMID 10523153
- [Background] Rice HE, Skinner MA, Mahaffey SM, Oldham KT, Ing RJ, Hale LP, Markert ML. Thymic transplantation for complete DiGeorge syndrome: medical and surgical considerations. J Pediatr Surg. 2004 Nov;39(11):1607-15. doi: 10.1016/j.jpedsurg.2004.07.020. PMID 15547821
- [Background] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Background] Albuquerque AS, Marques JG, Silva SL, Ligeiro D, Devlin BH, Dutrieux J, Cheynier R, Pignata C, Victorino RM, Markert ML, Sousa AE. Human FOXN1-deficiency is associated with alphabeta double-negative and FoxP3+ T-cell expansions that are distinctly modulated upon thymic transplantation. PLoS One. 2012;7(5):e37042. doi: 10.1371/journal.pone.0037042. Epub 2012 May 10. PMID 22590644
- [Background] Davies EG, Cheung M, Gilmour K, Maimaris J, Curry J, Furmanski A, Sebire N, Halliday N, Mengrelis K, Adams S, Bernatoniene J, Bremner R, Browning M, Devlin B, Erichsen HC, Gaspar HB, Hutchison L, Ip W, Ifversen M, Leahy TR, McCarthy E, Moshous D, Neuling K, Pac M, Papadopol A, Parsley KL, Poliani L, Ricciardelli I, Sansom DM, Voor T, Worth A, Crompton T, Markert ML, Thrasher AJ. Thymus transplantation for complete DiGeorge syndrome: European experience. J Allergy Clin Immunol. 2017 Dec;140(6):1660-1670.e16. doi: 10.1016/j.jaci.2017.03.020. Epub 2017 Apr 8. PMID 28400115
- [Background] Markert ML, Gupton SE, McCarthy EA. Experience with cultured thymus tissue in 105 children. J Allergy Clin Immunol. 2022 Feb;149(2):747-757. doi: 10.1016/j.jaci.2021.06.028. Epub 2021 Aug 4. PMID 34362576
- [Background] Kampinga J, Schuurman HJ, Pol GH, Bartels H, Broekhuizen R, Vaessen LM, Tielen FJ, Rozing J, Blaauw EH, Roser B, et al. Vascular thymus transplantation in rats. Technique, morphology, and function. Transplantation. 1990 Oct;50(4):669-78. doi: 10.1097/00007890-199010000-00028. PMID 2219290
- [Background] Jiang J, Wang H, Madrenas J, Zhong R. Surgical technique for vascularized thymus transplantation in mice. Microsurgery. 1999;19(2):56-60. doi: 10.1002/(sici)1098-2752(1999)19:23.0.co;2-f. PMID 10188826
- [Background] Ortak T, Oke R, Unsal M, Carnevale K, Siemionow M. A model of vascular thymus transplantation in athymic rats. Transplant Proc. 2001 Feb-Mar;33(1-2):372-4. doi: 10.1016/s0041-1345(00)02053-4. No abstract available. PMID 11266867
- [Background] LaMattina JC, Kumagai N, Barth RN, Yamamoto S, Kitamura H, Moran SG, Mezrich JD, Sachs DH, Yamada K. Vascularized thymic lobe transplantation in miniature swine: I. Vascularized thymic lobe allografts support thymopoiesis. Transplantation. 2002 Mar 15;73(5):826-31. doi: 10.1097/00007890-200203150-00032. PMID 11907438
- [Background] Zhao D, Qiu J, Wang C, Liu L, Li J, Chen L. Vascularized whole thymus transplantation in Rowett nude rats: effect of thymus allograft volume on tolerance induction. Transpl Immunol. 2010 May;23(1-2):40-4. doi: 10.1016/j.trim.2010.03.007. Epub 2010 Apr 1. PMID 20362672
- [Background] Zhao D, Wang L, Na N, Huang Z, Miao B, Hong L. A model of isolated, vascular whole thymus transplantation in nude rats. Transplant Proc. 2012 Jun;44(5):1394-8. doi: 10.1016/j.transproceed.2011.10.055. PMID 22664022
- [Background] Tintinago-Londono LF, Isaza-Pierotti DF, Restrepo JG, Rico-Sierra MJ, Osorio-Cardona JJ, Candelo E, Martinez FJ. Vascular Neonatal Thymus Transplantation in Rabbits. Transplant Proc. 2022 Oct;54(8):2381-2387. doi: 10.1016/j.transproceed.2022.08.035. Epub 2022 Oct 18. PMID 36270856
- [Background] MILLER JF. Role of the thymus in murine leukaemia. Nature. 1959 Apr 11;183(4667):1069. doi: 10.1038/1831069a0. No abstract available. PMID 13644292
- [Background] MILLER JF. Fate of subcutaneous thymus grafts in thymectomized mice inoculated with leukaemic filtrate. Nature. 1959 Dec 5;184(Suppl 23):1809-10. doi: 10.1038/1841809a0. No abstract available. PMID 14422530
- [Background] MILLER JF. Recovery of leukaemogenic agent from nonleukaemic tissues of thymectomized mice. Nature. 1960 Aug 20;187:703. doi: 10.1038/187703a0. No abstract available. PMID 14422531
- [Background] MILLER JF. Analysis of the thymus influence in leukaemogenesis. Nature. 1961 Jul 15;191:248-9. doi: 10.1038/191248a0. No abstract available. PMID 13770811
- [Background] MILLER JF. Etiology and pathogenesis of mouse leukemia. Adv Cancer Res. 1961;6:291-368. doi: 10.1016/s0065-230x(08)60623-5. No abstract available. PMID 14474037
- [Background] MILLER JF. Immunological function of the thymus. Lancet. 1961 Sep 30;2(7205):748-9. doi: 10.1016/s0140-6736(61)90693-6. No abstract available. PMID 14474038
- [Background] Miller A, Morse HC 3rd, Winkelstein J, Nathanson N. The role of antibody in recovery from experimental rabies. I. Effect of depletion of B and T cells. J Immunol. 1978 Jul;121(1):321-6. PMID 307577
- [Background] MCINTIRE KR, SELL S, MILLER JF. PATHOGENESIS OF THE POST-NEONATAL THYMECTOMY WASTING SYNDROME. Nature. 1964 Oct 10;204:151-5. doi: 10.1038/204151a0. No abstract available. PMID 14222260
- [Background] MILLER JF. INFLUENCE OF THYMECTOMY ON TUMOR INDUCTION BY POLYOMA VIRUS IN C57BL MICE. Proc Soc Exp Biol Med. 1964 Jun;116:323-7. doi: 10.3181/00379727-116-29237. No abstract available. PMID 14189129
- [Background] Mitchell GF, Miller JF. Immunological activity of thymus and thoracic-duct lymphocytes. Proc Natl Acad Sci U S A. 1968 Jan;59(1):296-303. doi: 10.1073/pnas.59.1.296. No abstract available. PMID 4873344
- [Background] Miller JF, Mitchell GF. Cell to cell interaction in the immune response. I. Hemolysin-forming cells in neonatally thymectomized mice reconstituted with thymus or thoracic duct lymphocytes. J Exp Med. 1968 Oct 1;128(4):801-20. doi: 10.1084/jem.128.4.801. PMID 5691985
- [Background] Mitchell GF, Miller JF. Cell to cell interaction in the immune response. II. The source of hemolysin-forming cells in irradiated mice given bone marrow and thymus or thoracic duct lymphocytes. J Exp Med. 1968 Oct 1;128(4):821-37. doi: 10.1084/jem.128.4.821. PMID 5691986
- [Background] Sprent J, Miller JF, Mitchell GF. Antigen-induced selective recruitment of circulating lymphocytes. 1971. J Immunol. 2006 Aug 1;177(3):1381-91. No abstract available. PMID 16849441
- [Background] Basten A, Miller JF, Sprent J, Pye J. A receptor for antibody on B lymphocytes. I. Method of detection and functional significance. J Exp Med. 1972 Mar 1;135(3):610-26. doi: 10.1084/jem.135.3.610. PMID 5058234
- [Background] Owens T, Fazekas de St Groth B, Miller JF. Coaggregation of the T-cell receptor with CD4 and other T-cell surface molecules enhances T-cell activation. Proc Natl Acad Sci U S A. 1987 Dec;84(24):9209-13. doi: 10.1073/pnas.84.24.9209. PMID 3501123
- [Background] Hoffmann MW, Allison J, Miller JF. Tolerance induction by thymic medullary epithelium. Proc Natl Acad Sci U S A. 1992 Apr 1;89(7):2526-30. doi: 10.1073/pnas.89.7.2526. PMID 1557355
- [Background] Miller JF. The golden anniversary of the thymus. Nat Rev Immunol. 2011 May 27;11(7):489-95. doi: 10.1038/nri2993. PMID 21617694
- [Background] Yan F, Mo X, Liu J, Ye S, Zeng X, Chen D. Thymic function in the regulation of T cells, and molecular mechanisms underlying the modulation of cytokines and stress signaling (Review). Mol Med Rep. 2017 Nov;16(5):7175-7184. doi: 10.3892/mmr.2017.7525. Epub 2017 Sep 19. PMID 28944829
- [Background] Gui J, Mustachio LM, Su DM, Craig RW. Thymus Size and Age-related Thymic Involution: Early Programming, Sexual Dimorphism, Progenitors and Stroma. Aging Dis. 2012 Jun;3(3):280-90. Epub 2012 Mar 14. PMID 22724086
- [Background] Appay V, Sauce D, Prelog M. The role of the thymus in immunosenescence: lessons from the study of thymectomized individuals. Aging (Albany NY). 2010 Mar 20;2(2):78-81. doi: 10.18632/aging.100122. PMID 20354268
- [Background] Griesemer AD, Sorenson EC, Hardy MA. The role of the thymus in tolerance. Transplantation. 2010 Sep 15;90(5):465-74. doi: 10.1097/TP.0b013e3181e7e54f. PMID 20555306
- [Background] Thapa P, Farber DL. The Role of the Thymus in the Immune Response. Thorac Surg Clin. 2019 May;29(2):123-131. doi: 10.1016/j.thorsurg.2018.12.001. Epub 2019 Mar 7. PMID 30927993
- [Background] Dukor P, Miller JF, House W, Allman V. Regeneration of thymus grafts. I. Histological and cytological aspects. Transplantation. 1965 Sep;3(5):639-68. doi: 10.1097/00007890-196509000-00006. No abstract available. PMID 5828539
- [Background] Gaugas JM, Rees RJ, Weddell AG, Palmer E. Reversal effect of thymus grafts on lepromatous leprosy in thymectomized-irradiated mice. Int J Lepr Other Mycobact Dis. 1971 Apr-Jun;39(2):388-95. No abstract available. PMID 5169805
- [Background] Marcolongo R, Di Paolo N. Fetal thymic transplant in patients with Hodgkin's disease. Blood. 1973 May;41(5):625-33. No abstract available. PMID 4694079
- [Background] Radov LA, Sussdorf DH, McCann RL. Relationship between age of allogeneic thymus donor and immunological restoration of athymic ('nude") mice. Immunology. 1975 Dec;29(6):977-88. PMID 1193689
- [Background] Hong R, Santosham M, Schulte-Wissermann H, Horowitz S, Hsu SH, Winkelstein JA. Reconstitution of B and T lymphocyte function in severe combined immunodeficiency disease after transplantation with thymic epithelium. Lancet. 1976 Dec 11;2(7998):1270-2. doi: 10.1016/s0140-6736(76)92031-6. PMID 63746
- [Background] Ballow M, Hyman LR. Combination immunotherapy in chronic mucocutaneous candidiasis. Synergism between transfer factor and fetal thymus tissue. Clin Immunol Immunopathol. 1977 Nov;8(3):504-12. doi: 10.1016/0090-1229(77)90014-9. No abstract available. PMID 912947
- [Background] Kindred B. Nude mice in immunology. Prog Allergy. 1979;26:137-238. No abstract available. PMID 386358
- [Background] Kaminski MJ, Ksiazek T. Vascularization of murine lymphoid tissue from various organs transplanted under the kidney capsule of syngeneic host. Acta Med Pol. 1980;21(3):219-26. No abstract available. PMID 6166151
- [Background] Zinkernagel RM. Restriction specificity of virus-specific cytotoxic T cells from thymectomised irradiated bone marrow chimeras reconstituted with thymus grafts. Thymus. 1981 Apr;2(6):321-7. PMID 6168044
- [Background] Ba D, Takeichi N, Kodama T, Kobayashi H. Restoration of T cell depression and suppression of blood pressure in spontaneously hypertensive rats (SHR) by thymus grafts or thymus extracts. J Immunol. 1982 Mar;128(3):1211-6. PMID 6120194
- [Background] Schuurman HJ, Vos JG, van de Brink E, Kater L. Culture of thymic epithelium for transplantation purposes: morphological characterization and in vivo biological effect on thymus-dependent immunity in athymic (nude) rats. Clin Immunol Immunopathol. 1982 Sep;24(3):418-31. doi: 10.1016/0090-1229(82)90012-5. No abstract available. PMID 6982141
- [Background] Atkinson K, Storb R, Ochs HD, Goehle S, Sullivan KM, Witherspoon RP, Lum LG, Tsoi MS, Sanders JE, Parr M, Stewart P, Thomas ED. Thymus transplantation after allogeneic bone marrow graft to prevent chronic graft-versus-host disease in humans. Transplantation. 1982 Feb;33(2):168-73. doi: 10.1097/00007890-198202000-00012. No abstract available. PMID 7036469
- [Background] Kast WM, de Waal LP, Melief CJ. Thymus dictates major histocompatibility complex (MHC) specificity and immune response gene phenotype of class II MHC-restricted T cells but not of class I MHC-restricted T cells. J Exp Med. 1984 Dec 1;160(6):1752-66. doi: 10.1084/jem.160.6.1752. PMID 6096476
- [Background] Ikehara S, Tanaka H, Nakamura T, Furukawa F, Inoue S, Sekita K, Shimizu J, Hamashima Y, Good RA. The influence of thymic abnormalities on the development of autoimmune diseases. Thymus. 1985;7(1):25-36. PMID 3871979
- [Background] Schuurman HJ, Vos JG, Broekhuizen R, Brandt CJ, Kater L. In vivo biological effect of allogeneic cultured thymic epithelium on thymus-dependent immunity in athymic nude rats. Scand J Immunol. 1985 Jan;21(1):21-30. doi: 10.1111/j.1365-3083.1985.tb01398.x. PMID 3871535
- [Background] Schuurman HJ, Vaessen LM, Vos JG, Hertogh A, Geertzema JG, Brandt CJ, Rozing J. Implantation of cultured thymic fragments in congenitally athymic nude rats: ignorance of thymic epithelial haplotype in generation of alloreactivity. J Immunol. 1986 Oct 15;137(8):2440-7. PMID 3760564
- [Background] Hong R. Reconstitution of T-cell deficiency by thymic hormone or thymus transplantation therapy. Clin Immunol Immunopathol. 1986 Jul;40(1):136-41. doi: 10.1016/0090-1229(86)90077-2. PMID 3521966
- [Background] Danner SA, Schuurman HJ, Lange JM, Gmelig Meyling FH, Schellekens PT, Huber J, Kater L. Implantation of cultured thymic fragments in patients with acquired immunodeficiency syndrome. Arch Intern Med. 1986 Jun;146(6):1133-6. PMID 2940985
- [Background] Dwyer JM, Wood CC, McNamara J, Kinder B. Transplantation of thymic tissue into patients with AIDS. An attempt to reconstitute the immune system. Arch Intern Med. 1987 Mar;147(3):513-7. PMID 3827429
- [Background] Touraine JL, Roncarolo MG, Royo C, Touraine F. Fetal tissue transplantation, bone marrow transplantation and prospective gene therapy in severe immunodeficiencies and enzyme deficiencies. Thymus. 1987;10(1-2):75-87. doi: 10.1007/978-94-009-3365-1_8. PMID 3324405
- [Background] Ohki H, Martin C, Corbel C, Coltey M, Le Douarin NM. Tolerance induced by thymic epithelial grafts in birds. Science. 1987 Aug 28;237(4818):1032-5. doi: 10.1126/science.3616623.
- [Background] Schuurman HJ, Vaessen LM, Broekhuizen R, Brandt CJ, Holewijn MC, Vos JG, Rozing J. Implantation of cultured thymic fragments in congenitally athymic (nude) rats. Influx of lymphocytes and dendritic cells. Scand J Immunol. 1987 Aug;26(2):129-39. doi: 10.1111/j.1365-3083.1987.tb02245.x. PMID 3498208
- [Background] Jotereau F, Heuze F, Salomon-Vie V, Gascan H. Cell kinetics in the fetal mouse thymus: precursor cell input, proliferation, and emigration. J Immunol. 1987 Feb 15;138(4):1026-30. PMID 2879866
- [Background] Georgiou HM, Lagarde AC, Bellgrau D. T cell dysfunction in the diabetes-prone BB rat. A role for thymic migrants that are not T cell precursors. J Exp Med. 1988 Jan 1;167(1):132-48. doi: 10.1084/jem.167.1.132. PMID 2961842
- [Background] McCune JM, Namikawa R, Kaneshima H, Shultz LD, Lieberman M, Weissman IL. The SCID-hu mouse: murine model for the analysis of human hematolymphoid differentiation and function. Science. 1988 Sep 23;241(4873):1632-9. doi: 10.1126/science.241.4873.1632. PMID 2971269
- [Background] Nikolic B, Gardner JP, Scadden DT, Arn JS, Sachs DH, Sykes M. Normal development in porcine thymus grafts and specific tolerance of human T cells to porcine donor MHC. J Immunol. 1999 Mar 15;162(6):3402-7. PMID 10092795
- [Background] Zhao Y, Sergio JJ, Swenson K, Arn JS, Sachs DH, Sykes M. Positive and negative selection of functional mouse CD4 cells by porcine MHC in pig thymus grafts. J Immunol. 1997 Sep 1;159(5):2100-7. PMID 9278295
- [Background] Yan Y, Devos T, Yu L, Xia G, Rutgeerts O, Goebels J, Segers C, Lin Y, Vandeputte M, Waer M. Pathogenesis of autoimmunity after xenogeneic thymus transplantation. J Immunol. 2003 Jun 15;170(12):5936-46. doi: 10.4049/jimmunol.170.12.5936. PMID 12794120
- [Background] Mendez-Ferrer S, Bonnet D, Steensma DP, Hasserjian RP, Ghobrial IM, Gribben JG, Andreeff M, Krause DS. Bone marrow niches in haematological malignancies. Nat Rev Cancer. 2020 May;20(5):285-298. doi: 10.1038/s41568-020-0245-2. Epub 2020 Feb 28. PMID 32112045
- [Background] Megias-Vericat JE, Ballesta-Lopez O, Barragan E, Martinez-Cuadron D, Montesinos P. Tyrosine kinase inhibitors for acute myeloid leukemia: A step toward disease control? Blood Rev. 2020 Nov;44:100675. doi: 10.1016/j.blre.2020.100675. Epub 2020 Mar 2. PMID 32147087
- [Background] Tabe Y, Konopleva M, Andreeff M. Fatty Acid Metabolism, Bone Marrow Adipocytes, and AML. Front Oncol. 2020 Feb 18;10:155. doi: 10.3389/fonc.2020.00155. eCollection 2020. PMID 32133293
- [Background] Venditti A, Gale RP, Buccisano F, Ossenkoppele G. Should persons with acute myeloid leukemia (AML) in 1st histological complete remission who are measurable residual disease (MRD) test positive receive an allotransplant? Leukemia. 2020 Apr;34(4):963-965. doi: 10.1038/s41375-020-0780-6. Epub 2020 Mar 4. No abstract available. PMID 32132654
- [Background] Paczulla AM, Rothfelder K, Raffel S, Konantz M, Steinbacher J, Wang H, Tandler C, Mbarga M, Schaefer T, Falcone M, Nievergall E, Dorfel D, Hanns P, Passweg JR, Lutz C, Schwaller J, Zeiser R, Blazar BR, Caligiuri MA, Dirnhofer S, Lundberg P, Kanz L, Quintanilla-Martinez L, Steinle A, Trumpp A, Salih HR, Lengerke C. Absence of NKG2D ligands defines leukaemia stem cells and mediates their immune evasion. Nature. 2019 Aug;572(7768):254-259. doi: 10.1038/s41586-019-1410-1. Epub 2019 Jul 17. PMID 31316209
- [Background] Han Y, Dong Y, Yang Q, Xu W, Jiang S, Yu Z, Yu K, Zhang S. Acute Myeloid Leukemia Cells Express ICOS Ligand to Promote the Expansion of Regulatory T Cells. Front Immunol. 2018 Sep 26;9:2227. doi: 10.3389/fimmu.2018.02227. eCollection 2018. PMID 30319662
- [Background] Pohlenz P, Klatt J, Schon G, Blessmann M, Li L, Schmelzle R. Microvascular free flaps in head and neck surgery: complications and outcome of 1000 flaps. Int J Oral Maxillofac Surg. 2012 Jun;41(6):739-43. doi: 10.1016/j.ijom.2012.02.012. Epub 2012 Mar 17. PMID 22424757
- [Background] McCaughtry TM, Wilken MS, Hogquist KA. Thymic emigration revisited. J Exp Med. 2007 Oct 29;204(11):2513-20. doi: 10.1084/jem.20070601. Epub 2007 Oct 1. PMID 17908937
- [Background] Yamada K, Vagefi PA, Utsugi R, Kitamura H, Barth RN, LaMattina JC, Sachs DH. Thymic transplantation in miniature swine: III. Induction of tolerance by transplantation of composite thymokidneys across fully major histocompatibility complex-mismatched barriers. Transplantation. 2003 Aug 15;76(3):530-6. doi: 10.1097/01.TP.0000080608.42480.E8. PMID 12923439
- [Background] Valcarcel D, Sierra J, Wang T, Kan F, Gupta V, Hale GA, Marks DI, McCarthy PL, Oudshoorn M, Petersdorf EW, Ringden O, Setterholm M, Spellman SR, Waller EK, Gajewski JL, Marino SR, Senitzer D, Lee SJ. One-antigen mismatched related versus HLA-matched unrelated donor hematopoietic stem cell transplantation in adults with acute leukemia: Center for International Blood and Marrow Transplant Research results in the era of molecular HLA typing. Biol Blood Marrow Transplant. 2011 May;17(5):640-8. doi: 10.1016/j.bbmt.2010.07.022. Epub 2010 Jul 30. PMID 20674756
- [Background] Sanz J, Jaramillo FJ, Planelles D, Montesinos P, Lorenzo I, Moscardo F, Martin G, Lopez F, Martinez J, Jarque I, de la Rubia J, Larrea L, Sanz MA, Sanz GF. Impact on outcomes of human leukocyte antigen matching by allele-level typing in adults with acute myeloid leukemia undergoing umbilical cord blood transplantation. Biol Blood Marrow Transplant. 2014 Jan;20(1):106-10. PMID 24516896
- [Background] Shichkin VP, Antica M. Thymus Regeneration and Future Challenges. Stem Cell Rev Rep. 2020 Apr;16(2):239-250. doi: 10.1007/s12015-020-09955-y. PMID 31997162
- [Background] Ma L, Fei B. Comprehensive review of surgical microscopes: technology development and medical applications. J Biomed Opt. 2021 Jan;26(1):010901. doi: 10.1117/1.JBO.26.1.010901. PMID 33398948
- [Background] Tamai S. History of microsurgery. Plast Reconstr Surg. 2009 Dec;124(6 Suppl):e282-e294. doi: 10.1097/PRS.0b013e3181bf825e. PMID 19952697
- [Background] Badash I, Gould DJ, Patel KM. Supermicrosurgery: History, Applications, Training and the Future. Front Surg. 2018 Mar 21;5:23. doi: 10.3389/fsurg.2018.00023. eCollection 2018. PMID 29740586